CLINICAL TRIAL: NCT04632095
Title: Parasternal vs. Sternotomy Approach for Conventional Aortic Valve Replacement
Acronym: PASTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jena University Hospital (Other)
Collaborators: The German Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PASTA-UKJ
Record Dates: First submitted 2020-11-06; First posted 2020-11-17 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2020-11

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic Valve Stenosis; minimally invasive surgery; parasternal approach; quality of life; aortic valve replacement; inflammatory markers
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sternotomy AVR (Active Comparator): Aortic valve replacement due to sternotomy
  Interventions: Procedure: Aortic valve replacement due to sternotomy
- Mini AVR (Active Comparator): Aortic valve replacement due to parasternal right anterior mini-thoracotomy
  Interventions: Procedure: Aortic valve replacement due to parasternal right anterior mini-thoracotomy

INTERVENTIONS:
Procedure: Aortic valve replacement due to sternotomy — conventional surgery of aortic stenosis
  Arms: Sternotomy AVR
Procedure: Aortic valve replacement due to parasternal right anterior mini-thoracotomy — surgery of aortic stenosis in minimally invasive technique
  Arms: Mini AVR

SUMMARY:
Prospective randomized study comparing aortic valve replacement using parasternal or sternotomy access with regard to quality of life and systemic inflammatory reaction.

DETAILED DESCRIPTION:
The classic surgical treatment of aortic stenosis is valve replacement through complete midline opening of the breastbone (median sternotomy) and use of cardiopulmonary bypass (CPB). Risks of this procedure are related to both the surgical approach and the use of CPB. Using minimally invasive approaches in non-cardiac patients (e.g laparoscopy) resulted in reduced postoperative inflammatory response when compared to patients undergoing the same procedures carried out with a conventional "open" technique. Minimally invasive surgical approaches in which the sternum is partially opened (partial sternotomy) or not opened at all (parasternal access) have thus far shown similar procedure related mortality and lower incidence of perioperative complications, despite longer CPB times. Our single center experience thus far suggests superiority of parasternal aortic valve replacement (O/E ratio of 0.19 over the last 2 years), as well as a reduced postoperative inflammatory response (as measured by lower CRP (C reactive protein ) levels taken 6 hours post-surgery). However, these data have several confounders and there is currently no prospective randomized trial addressing this topic. We therefore conduct a randomized comparison of parasternal versus classic sternotomy aortic valve replacement. Based on our previous experience, we expect very low mortality risk in both groups (expected ≤ 1%). The primary endpoint is therefore quality of life assessed using the SF-36 (Short Form) health survey questionnaire. This approach is similar to other current large multicenter trials. In order to address the impact of reduced surgical trauma on inflammatory response; we will quantify an established panel of inflammatory markers (PCT, CRP, interleukin 6) and use bio-banking to allow for further in depth analysis later on. Standardized clinical endpoints will be analyzed as additional secondary parameters. Power analysis determined a number of 50 patients allocated to 2 equal groups to achieve a power of 80%. The parasternal approach is expected to be superior when compared to sternotomy in both the primary and some, if not most, secondary endpoints. We expect our study to become an important milestone for decision-making in the treatment of aortic stenosis. Patients currently fear sternotomy, but the less invasive transcatheter valve implantation appears to be limited by inferior long-term outcome. The parasternal, sternotomy-sparing, classic aortic valve replacement is therefore an attractive therapeutic alternative. Our investigation in relation to systemic inflammatory response will further shed light on the underlying mechanisms explaining differences in clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Indication for elective isolated aortic valve replacement
* Anatomical suitability for both sternotomy and parasternal access
* Age ≥ 18
* Written informed consent in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Planned simultaneous cardiac surgery interventions (Mitral valve surgery, tricuspid valve surgery, CABG, Pacemaker or defibrillator implantation, Pulmonalvenenisolation, Maze, closure of left atrial appendage , patent foramen ovale or atrial septal defect closure)
* Acute myocardial infarction within 4 weeks, coronary heart disease
* Acute endocarditis
* TIA or stroke within 6 months prior to the procedure
* Pregnant or breast-feeding women
* Renal failure requiring dialysis
* Ejection fraction ≤ 30%
* Re-operation
* Disease with a life expectancy < 2 years
* Therapy with glucocorticoids or immunosuppressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-03-16 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
Quality of life - physical function | 30 days after surgery
  Comparison of the physical quality of life between the two groups 30 days after surgery using the physical function score of the 36-Item Short Form Health Survey (SF-36). The physical function score is a scale from 0 (poor physical function) to 100 (excellent physical function, with an average score of 50. It includes items that assess physical functioning, bodily pain, physical role functioning, vitality, and generaly health perceptions.

SECONDARY OUTCOMES:
Inflammatory markers: Procalcitonin, C-reactive protein, Interleukin-6 | During the first 48 hours after surgery
  Plasma profiles of inflammatory biomarkers at defined time points in the course of the surgical intervention (baseline, before introduction of CPB, 1 hour after introduction of CPB, disconnection of CPB, 6, 24 and 48 hours post-surgery)
Quality of Life - mental function | 30 days after surgery
  Comparison of the mental quality of life between the two Groups 30 days after surgery using the mental component score of the 36-Item Short Form Health Survey (SF-36). The mental function score is a scale from 0 (poor mental quality of life) to 100 (excellent mental quality of life), with an average score of 50. It includes items that assess vitality, general health perceptions, emotional role functioning, social role functioning, and mental health.
Duration of the Operation | During the aortic valve replacement surgery
  Comparison of the average duration of operation between the groups
Duration of cardiopulmonary bypass | During the aortic valve replacement surgery
  Comparison of the average duration of cardiopulmonary bypass between the groups
Duration of aortic clamping | During the aortic valve replacement surgery
  Comparison of the average duration of aortic clamping between the two groups
Major Adverse Cardiac and Cerebrovascular Events (MACCE) | From the time of surgery until the patient is discharged from hospital, an average of 7 days
  A composite endpoint of mortality, myocardial infarction, urgent revascularization, stroke and major bleeding
Blood transfusion | From the time of surgery until the patient is discharged from hospital, an average of 7 days
  A comparison of the number of transfusions between the groups
Rethoracotomy for bleeding | From the time of surgery until the patient is discharged from hospital, an average of 7 days
  The incidence of rethoracotomy for bleeding after surgery
Post-operative pain | From the time of surgery until the patient is discharged from hospital, an average of 7 days
  Measurement of patient's subjective assessment of their pain after surgery using a visual scale
Duration of mechanical ventilation | Measured from the time of arrival in the Intensive Care Unit until the time patients are extubated, an average of 12 hours
  Comparison of the average duration of mechanical ventilation between the groups
Length of ICU stay | From the time of surgery until the patient is discharged from hospital, an average of 30 days
  Comparison of the average number of days spent in Intensive Care Unit between the two groups
Length of hospital stay | From the time of surgery until the patient is discharged from hospital, an average of 30 days
  Comparison of the average number of days spent in hospital between the groups
Atrial fibrillation | From the time of surgery until the patient is discharged from hospital, an average of 7 days
  Incidence of new-onset atrial fibrillation after cardiac surgery
Wound infection | During the first 30 days after surgery
  Incidence of wound infections
Mortality | During the first 30 days after surgery
  intra- and postoperative mortality

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Tkebuchava, MD, Principal Investigator — University Hospital Jena; Torsten Doenst, MD, Principal Investigator — University Hospital Jena
Locations (1):
- UKJ, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No